CLINICAL TRIAL: NCT02447536
Title: Evaluating the Effect of Different BCG Strains on Early Life Hospital Admissions in Guinea-Bissau: A Randomised Trial
Brief Title: Trial of Two Strains of BCG
Acronym: BCGSTRAIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BCGSTRAIN
Record Dates: First submitted 2015-04-20; First posted 2015-05-19 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Morbidity; Bacille Calmette-Guérin
Keywords: Immunization; Morbidity; Mortality; BCG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BCG-DENMARK (Active Comparator): Infants randomised to receive BCG-DENMARK at dismissal from the Maternity Ward will receive one 0.05 ml dose of Mycobacterium bovis BCG live attenuated vaccine BCG-Denmark 1331 (Statens Serum Institute) by intradermal injection in the left deltoid region. Dependent on national supply, infants will receive oral polio vaccine (OPV) at the time of BCG-vaccination.
  NOTE: By 1st of July 2016, infants in this arm has received BCG-Japan due to a worldwide shortage of BCG-Denmark because of a halt in production of this vaccine at the Statens Serum Institut in Copenhagen.
  Interventions: Biological: BCG-Denmark 1331 (Statens Serum Institute)
- BCG-RUSSIA (Active Comparator): Infants randomised to receive BCG-RUSSIA at dismissal from the Maternity Ward will receive one 0.05 ml dose Mycobacterium bovis BCG live attenuated vaccine BCG-Russia-I (Serum Institute of India) by intradermal injection in the left deltoid region. Dependent on national supply, infants will receive oral polio vaccine (OPV) at the time of BCG-vaccination.
  Interventions: Biological: BCG-Russia-I (Serum Institute of India)

INTERVENTIONS:
Biological: BCG-Denmark 1331 (Statens Serum Institute) — See above
  Arms: BCG-DENMARK
Biological: BCG-Russia-I (Serum Institute of India) — See above
  Arms: BCG-RUSSIA

SUMMARY:
The investigators aim to conduct a randomised controlled trial comparing two Bacille Calmette-Guérin (BCG) strains currently used in Guinea-Bissau, the Danish and the Russian, in terms of prevention of neonatal and early life morbidity and mortality, immune responses and adverse events related to BCG vaccination. The primary outcome will be hospital admissions within 6 weeks of age.

DETAILED DESCRIPTION:
BACKGROUND At the Bandim Health Project (www.bandim.org) in Guinea-Bissau, we observed that Bacille Calmette-Guérin (BCG) vaccination at birth is associated with survival benefits which cannot be explained by prevention of tuberculosis (TB), which is rare during the first year of life. There is mounting evidence that the beneficial effects of BCG on neonatal mortality stems from non-specific beneficial immune training, also termed heterologous immunity. This way, BCG immunisation possibly confers enhanced protection against a broad range of severe infections such as pneumonia and septicemia.

In addition, observational studies from Guinea-Bissau suggest that BCG-vaccinated children who produced a scar upon immunisation have significantly better survival than BCG-vaccinated children who did not produce a scar. The pattern is the same with regard to PPD (tuberculin) skin test. While correct BCG-vaccination technique is undoubtedly important for scarring, several studies have shown that the strain of BCG might be important as well.

Globally, BCG coverage exceeds 90%, making BCG the most widely used vaccine in the world. According to UNICEF, the annual demand for the BCG vaccine was 130 million doses in 2013. Several different vaccine strains are being used, yet few studies have compared the different strains. However, several animal and human studies have shown that these genetically diverse vaccine strains induce different protective efficacy against TB, risk of adverse events and susceptibility to anti-TB drugs. Recently, a large observational study based in Uganda showed that there were significant differences between BCG strains concerning the response to specific mycobacteria and non-specific immune responses. In particular, BCG-Denmark was associated with a much higher rate of scarring (93%) than BCG-Russia (52%), but also a higher rate of adverse events in terms of ulcers and abscesses (1.8% versus 0.3%).

OBJECTIVE We aim to compare the effect of two strains of BCG (BCG-Denmark, BCG-Russia) provided at birth to children born at the National Hospital Simão Mendes (HNSM) on subsequent hospitalisations. Furthermore, mortality in the first 6 weeks and adverse events at 2 and 6 months of age will be reported for all children, and BCG scar frequency (2 and 6 months) and PPD response (6 months) will be reported for a proportion of the infants.

METHODS The study will be conducted by the Bandim Health Project (BHP). The BHP maintains a health and demographic surveillance system (HDSS) in 6 districts of the capital in Guinea-Bissau covering approximately 102,000 inhabitants. All houses in the HDSS are visited monthly and all pregnancies and births are registered.

Study participants will be enrolled at the National Hospital and followed up through the HDSS and by telephone interviews as well as through hospital records. The study will be individually randomised, with 1:1 randomisation between the two strains (BCG-Denmark, BCG-Russia). During a two year inclusion period, we expect to be able to include at least 12,000 children, i.e. 6,000 in each BCG strain group. Of these, around 25% will reside within the HDSS.

ELIGIBILITY:
Inclusion Criteria:

Newborn infants at the HNSM maternity ward.

Exclusion Criteria:

Infants included in another randomized trial of BCG. Infants with a severe congenital abnormality.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12006 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-11-24 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Hospital admission | 6 weeks after birth

SECONDARY OUTCOMES:
Mortality | 6 weeks
  Reported exclusively for a subgroup of infants with regular house visits
BCG scar frequency | 6 months
  Reported exclusively for a subgroup of infants with regular house visits
PPD (tuberculin response) | 6 months
  Reported exclusively for a subgroup of infants with regular house visits
Adverse events (abscesses/ulcers) | 6 months
  Adverse events to the vaccines will be evaluated for a subgroup of infants with regular house visits
Hospital admission during neonatal period | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Aaby, Prof., Principal Investigator — Bandim Health Project
Locations (1):
- Bandim Health Project, Apartado 861, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wardlaw T, You D, Newby H, Anthony D, Chopra M. Child survival: a message of hope but a call for renewed commitment in UNICEF report. Reprod Health. 2013 Dec 11;10:64. doi: 10.1186/1742-4755-10-64. PMID 24325885
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] Penfold S, Willey BA, Schellenberg J. Newborn care behaviours and neonatal survival: evidence from sub-Saharan Africa. Trop Med Int Health. 2013 Nov;18(11):1294-316. doi: 10.1111/tmi.12193. Epub 2013 Sep 24. PMID 24112377
- [Background] Aaby P, Roth A, Ravn H, Napirna BM, Rodrigues A, Lisse IM, Stensballe L, Diness BR, Lausch KR, Lund N, Biering-Sorensen S, Whittle H, Benn CS. Randomized trial of BCG vaccination at birth to low-birth-weight children: beneficial nonspecific effects in the neonatal period? J Infect Dis. 2011 Jul 15;204(2):245-52. doi: 10.1093/infdis/jir240. PMID 21673035
- [Background] Biering-Sorensen S, Aaby P, Napirna BM, Roth A, Ravn H, Rodrigues A, Whittle H, Benn CS. Small randomized trial among low-birth-weight children receiving bacillus Calmette-Guerin vaccination at first health center contact. Pediatr Infect Dis J. 2012 Mar;31(3):306-8. doi: 10.1097/INF.0b013e3182458289. PMID 22189537
- [Background] Roth A, Gustafson P, Nhaga A, Djana Q, Poulsen A, Garly ML, Jensen H, Sodemann M, Rodriques A, Aaby P. BCG vaccination scar associated with better childhood survival in Guinea-Bissau. Int J Epidemiol. 2005 Jun;34(3):540-7. doi: 10.1093/ije/dyh392. Epub 2005 Jan 19. PMID 15659474
- [Background] Garly ML, Martins CL, Bale C, Balde MA, Hedegaard KL, Gustafson P, Lisse IM, Whittle HC, Aaby P. BCG scar and positive tuberculin reaction associated with reduced child mortality in West Africa. A non-specific beneficial effect of BCG? Vaccine. 2003 Jun 20;21(21-22):2782-90. doi: 10.1016/s0264-410x(03)00181-6. PMID 12798618
- [Background] Roth A, Sodemann M, Jensen H, Poulsen A, Gustafson P, Weise C, Gomes J, Djana Q, Jakobsen M, Garly ML, Rodrigues A, Aaby P. Tuberculin reaction, BCG scar, and lower female mortality. Epidemiology. 2006 Sep;17(5):562-8. doi: 10.1097/01.ede.0000231546.14749.ab. PMID 16878042
- [Background] Behr MA. BCG--different strains, different vaccines? Lancet Infect Dis. 2002 Feb;2(2):86-92. doi: 10.1016/s1473-3099(02)00182-2. PMID 11901655
- [Background] Ritz N, Curtis N. Mapping the global use of different BCG vaccine strains. Tuberculosis (Edinb). 2009 Jul;89(4):248-51. doi: 10.1016/j.tube.2009.03.002. Epub 2009 Jun 18. PMID 19540166
- [Background] Behr MA. Correlation between BCG genomics and protective efficacy. Scand J Infect Dis. 2001;33(4):249-52. doi: 10.1080/003655401300077180. PMID 11345214
- [Background] Ritz N, Hanekom WA, Robins-Browne R, Britton WJ, Curtis N. Influence of BCG vaccine strain on the immune response and protection against tuberculosis. FEMS Microbiol Rev. 2008 Aug;32(5):821-41. doi: 10.1111/j.1574-6976.2008.00118.x. Epub 2008 Jul 9. PMID 18616602
- [Background] Anderson EJ, Webb EL, Mawa PA, Kizza M, Lyadda N, Nampijja M, Elliott AM. The influence of BCG vaccine strain on mycobacteria-specific and non-specific immune responses in a prospective cohort of infants in Uganda. Vaccine. 2012 Mar 9;30(12):2083-9. doi: 10.1016/j.vaccine.2012.01.053. Epub 2012 Jan 31. PMID 22300718
- [Background] Biai S, Rodrigues A, Nielsen J, Sodemann M, Aaby P. Vaccination status and sequence of vaccinations as risk factors for hospitalisation among outpatients in a high mortality country. Vaccine. 2011 May 9;29(20):3662-9. doi: 10.1016/j.vaccine.2011.03.016. Epub 2011 Apr 6. PMID 21440640
- [Background] Aaby P, Whittle H, Benn CS. Vaccine programmes must consider their effect on general resistance. BMJ. 2012 Jun 14;344:e3769. doi: 10.1136/bmj.e3769. No abstract available. PMID 22700785
- [Result] Schaltz-Buchholzer F, Bjerregaard-Andersen M, Oland CB, Golding C, Stjernholm EB, Monteiro I, Aaby P, Benn CS. Early Vaccination With Bacille Calmette-Guerin-Denmark or BCG-Japan Versus BCG-Russia to Healthy Newborns in Guinea-Bissau: A Randomized Controlled Trial. Clin Infect Dis. 2020 Nov 5;71(8):1883-1893. doi: 10.1093/cid/ciz1080. PMID 31677386
- [Derived] Schaltz-Buchholzer F, Bjerregard Oland C, Berendsen M, Bjerregaard-Andersen M, Stjernholm EB, Golding CN, Monteiro I, Aaby P, Benn CS. Maternal BCG primes for enhanced health benefits in the newborn. J Infect. 2022 Mar;84(3):321-328. doi: 10.1016/j.jinf.2021.12.028. Epub 2021 Dec 24. PMID 34958808
- [Derived] Schaltz-Buchholzer F, Berendsen M, Roth A, Jensen KJ, Bjerregaard-Andersen M, Kjaer Sorensen M, Monteiro I, Aaby P, Stabell Benn C. BCG skin reactions by 2 months of age are associated with better survival in infancy: a prospective observational study from Guinea-Bissau. BMJ Glob Health. 2020 Sep;5(9):e002993. doi: 10.1136/bmjgh-2020-002993. PMID 32978212